CLINICAL TRIAL: NCT00670527
Title: Evaluation of [18F] Fluorocholine PET/CT for Detection of Regional Lymph Node Metastases From Prostate Cancer
Brief Title: [18F] Fluorocholine FCH Positron Emission Tomography (PET)/Computed Tomography (CT) for Detection of Prostate Cancer Lymph Nodes Metastases
Acronym: PROPET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Mads Hvid Poulsen, MD, Department of Urology, Odense University Hospital, Denmark
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: PROPET, Project nr. 104.
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; [18F] Fluorocholine PET/CT; FCH; lymph node metastasis; staging; sensitivity; specificity; PROPET
MeSH Terms: conditions — Prostatic Neoplasms; Lymphatic Metastasis; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: [18F] Fluorocholine PET/CT — The patients fast 6 hours before the [18F]Fluorocholine PET/CT scan. [18F]Fluorocholine will be used as tracer with a dosage of 4 MBq per kg bodyweight. PET/CT imaging will be performed after 15 and 60 after the intravenous injection of the tracer. The patient will receive 2 full body FCH PET/CT. The CT scan is with contrast.
  The radiation exposure from the CT scan is 9 mSv and from the PET scan it is 3 mSv, giving a total of 12 mSv, which equals 4 times the yearly background radiation in Denmark.

SUMMARY:
The objective of this trial is to assess the value of 18F-choline PET/CT for the detection of regional lymph node metastases from prostate cancer. In addition, the investigators want to evaluate whether 18F-choline PET/CT can replace lymphadenectomy for the staging of prostate cancer.

DETAILED DESCRIPTION:
The purpose of this prospective trail is to improve the staging of patients with prostate cancer. The investigators focus on the group of patients with a newly diagnosed prostate cancer, and specifically the ones who have an intermediate and high risk of disseminated prostate cancer.

The aim is to improve staging by replacing the traditional invasive method, the lymphadenectomy, which has a rather low sensitivity by a non-invasive method, 18F-choline PET/CT which has a presumably superior sensitivity.

The treatment of patients with prostate cancer relies on the stage of the disease. Patients with disseminated prostate cancer are incurable and are treated with palliatively. In contrast, patients with localized prostate cancer are offered curative therapy. Hence, the stage of prostate cancer is crucial for the choice of treatment.

The potential benefits are

* The patients avoid the surgical trauma including complications and convalescents period.
* The accuracy of the prostate cancer staging is improved, the potential of which is better survival.

The patients are 18F-choline PET/CT scanned prior to their lymphadenectomy, the results of the 18F-choline PET/CT are blinded for the surgeon. The endpoint of the trail is the comparison of 18F-choline PET/CT and the histopathological investigation of the regional lymph nodes of prostate.

Assuming a prevalence of metastasised prostate cancer of 20% and a true (unknown) sensitivity of FCH PET/CT of 95%, 205 patients are sufficient to show that the sensitivity of the FCH PET/CT is greater than 80% with a power of 80% at significance level 5%. The size of the confidence interval for specificity of FCH PET/CT is expected to become reasonable small. In opposition to lymphadenectomy, FCH PET/CT results may point to metastases in neighbouring regions which gives an additional benefit to FCH PET/CT justifying a test level for sensitivity of 80%."

Accordingly 205 patients will be included over 2½ years. The first patients have been included in January 2008. Interim analyses will be done after 25, 50 and 100 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a biopsy confirmed prostate cancer who awaits curative treatment and have
* An elevated level of prostate-specific antigen PSA>10 ng/mL (nanogram per milliliter) or/and
* A Gleason score > 6 or/and
* A TNM staging of T3

Exclusion Criteria:

* Patients who withdraw their informed consent.
* Patients who have a bone scan indicates metastatic prostate cancer.
* Patients who have a TNM stage is T4

In the case we detect a patient having an obvious other major illness e.g. lung cancer, the patient is referred to relevant treatment. Depending on the illness the might be excluded from the study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2008-01; Primary Completion 2013-02 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
The primary target variable "metastasizes to regional lymph nodes" (yes/no) will be used to estimate the diagnostic usefulness of FCH PET/CT in terms of sensitivity, specificity, positive and negative predictive values. | The [18F] Fluorocholin PET/CT and the lymphadenectomi is done within 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Mads Hvid Poulsen, MD, Principal Investigator — Department of Urology, Odense University Hospital, Denmark; Ulla Geertsen, MD, Head of Department, Study Chair — Department of Urology, Odense University Hospital, Denmark; Niels Svolgaard, MD, Senior Physician, Study Chair — Department of Urology, Odense University Hospital, Denmark; Steen Walter, MD, DMSci, Professor, Study Chair — Department of Urology, Odense University Hospital, Denmark; Kirsten Bouchelouche, MD, DMSci, Study Chair — Odense University Hospital; Mette Høilund-Carlsen, Head Technician, Study Chair — Odense University Hospital; Henrik Petersen, MD, Senior Physician, Study Chair — Odense University Hospital; Mattias Ögren, Radiochemist, PhD, Study Chair — Odense University Hospital; Poul F Høilund-Carlsen, MD, DMSci, Professor, Study Chair — Department of Nuclear Medicine, Odense University Hospital, Demnark; Oke Gerke, Post-Doc, PhD, Study Chair — University of Southern Denmark; Werner Vach, PhD, Professor, Study Chair — University of Southern Denmark; Birgitte Svolgaard, MD, Senior Physician, Study Chair — Odense University Hospital; Niels Marcussen, MD, DMSci, Professor, Study Chair — Odense University Hospital
Locations (1):
- Department of Urology, Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Poulsen MH, Bouchelouche K, Hoilund-Carlsen PF, Petersen H, Gerke O, Steffansen SI, Marcussen N, Svolgaard N, Vach W, Geertsen U, Walter S. [18F]fluoromethylcholine (FCH) positron emission tomography/computed tomography (PET/CT) for lymph node staging of prostate cancer: a prospective study of 210 patients. BJU Int. 2012 Dec;110(11):1666-71. doi: 10.1111/j.1464-410X.2012.11150.x. Epub 2012 Apr 23. PMID 22520686